CLINICAL TRIAL: NCT07177222
Title: Quality of Life in Patients With Achalasia Cardia Before and After Esophagocardiomyotomy
Brief Title: Compare the Quality of Life of Patients With Achalasia Cardia (AC) After Laparoscopic and Open Esophagocardiomyotomy.
Acronym: GERD-HRQL
Status: Completed | Type: Observational
Sponsor: Osh State University (Other)
Collaborators: Kyrgyz State Medical Academy (Other)
Responsible Party: Principal Investigator, Zhypargul Abdullaeva, PhD, Osh State University
Other Study IDs: Quality of life in patients
Record Dates: First submitted 2025-08-29; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-07

CONDITIONS: Achalasia Cardia; GERD-HRQL Scale; Eckardt Scale
MeSH Terms: conditions — Esophageal Achalasia | interventions — Conversion to Open Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- 18 patients: underwent laparoscopic esophagocardiomyotomy
  Interventions: Procedure: laparoscopic esophagocardiomyotomy
- 20 patients: underwent open surgery
  Interventions: Procedure: open surgery

INTERVENTIONS:
Procedure: laparoscopic esophagocardiomyotomy — Heller myotomy, is a minimally invasive surgical procedure that involves cutting the muscle at the lower end of the esophagus to treat achalasia, a condition where this muscle (esophageal sphincter) fails to relax and hinders food passage into the stomach.
  Groups: 18 patients
Procedure: open surgery — Open surgery, or traditional surgery, involves a surgeon making one large incision to directly access and view the internal organ or body part being operated on.
  Groups: 20 patients

SUMMARY:
Study design. A randomized, prospective design study with retrospective data addition was conducted at two medical institutions between December 2017 and July 2025. Patients were equally allocated (1:1) between the laparoscopic and open Heller esophagocardiomyotomy groups.

Ethical aspects. All research procedures were carried out in accordance with the principles of the Helsinki Declaration and national ethical standards. The study protocol was approved by the Bioethics Committee of the Kyrgyz State Medical Academy (KSMA) named after I.K. Akhunbaev (protocol No. 6, dated 11.12.2017).

All participants were provided with a full explanation of the study objectives, methods, potential risks and benefits, and provided written informed consent prior to surgery and the processing of their anonymised clinical data for scientific purposes.

The study included 38 patients diagnosed with AC. The patients were divided into two groups: 18 patients underwent laparoscopic esophagocardiomyotomy, and 20 patients underwent open surgery.

A comparative analysis of these groups made it possible to evaluate the effectiveness and safety of both laparoscopic and traditional surgical interventions in the early and late postoperative periods.

All participants were provided with a full explanation of the study objectives, methods, potential risks and benefits, and provided written informed consent prior to surgery and the processing of their anonymised clinical data for scientific purposes.

The study included 38 patients diagnosed with AC. The patients were divided into two groups: 18 patients underwent laparoscopic esophagocardiomyotomy, and 20 patients underwent open surgery.

A comparative analysis of these groups made it possible to evaluate the effectiveness and safety of both laparoscopic and traditional surgical interventions in the early and late postoperative periods.

Inclusion criteria: Patients meeting the following requirements were accepted into the study:

* Clinically and instrumentally confirmed diagnosis of grade II-III AС, established on the basis of esophagogastroduodenoscopy, fluoroscopy with a contrast agent.
* No previous surgical operations on the esophagus and cardia;
* Availability of written informed consent for participation in the study and subsequent observation.

Exclusion criteria: Patients were excluded from the study if they had:

* Severe concomitant diseases (cardiovascular, respiratory, endocrine and others) that could limit the possibility of safe surgery and/or long-term observation;
* Detected malignant neoplasms of the esophagus, cardia or stomach;
* Refusal to participate in the study or inability to comply with the observation protocol. Preoperative preparation: All patients underwent a preoperative examination, which included: - Clinical history collection with a detailed description of complaints, duration and dynamics of the disease, presence of complications and concomitant diseases;
* General clinical and biochemical tests, electrocardiography;
* Esophagogastroduodenoscopy (EGDS) to assess the degree of expansion of the esophagus, the condition of the mucous membrane and to exclude tumor processes;
* X-ray examination of the esophagus with barium contrast to assess the degree of esophageal dilation, the functional state of the cardia and the identification of associated changes (diverticula, gastroesophageal reflux).

Surgical intervention. Classical esophagocardiomyotomy performed via laparotomy remains the accepted method of treating AC. The operation involves esophagocardiomyotomy using the Heller technique, which improves the passage of food and reduces swallowing difficulties and reflux of gastric contents.

Traditional laparotomy access is associated with high trauma and a long recovery period. Laparoscopic esophagocardiomyotomy in our study was performed using modern minimally invasive technologies.

ELIGIBILITY:
Inclusion Criteria:

* Clinically and instrumentally confirmed diagnosis of grade II-III AС, established based on esophagogastroduodenoscopy, fluoroscopy with a contrast agent;
* No previous surgical operations on the esophagus and cardia;
* Availability of written informed consent for participation in the study and subsequent observation.

Exclusion Criteria:

* Severe concomitant diseases (cardiovascular, respiratory, endocrine and others) that could limit the possibility of safe surgery and/or long-term observation;
* Detected malignant neoplasms of the esophagus, cardia or stomach;
* Refusal to participate in the study or inability to comply with the observation protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study included 38 patients diagnosed with AC. The patients were divided into two groups: 18 patients underwent laparoscopic esophagocardiomyotomy, and 20 patients underwent open surgery.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Significant and long-lasting reduction in symptom severity according to the Eckardt scale | from 6 to 60 months
  The patient's Eckardt score drops from a high value (indicating severe achalasia symptoms) to a low value (typically ≤3) and remains low over several years.

CONTACTS AND LOCATIONS:
Overall Officials: Bakytbek Osmonaliev, PhD, Principal Investigator — Kyrgyz State Medical Academy
Locations (1):
- Laparoscopic esophagocardiomyotomy, Bishkek, Kyrgyzstan